CLINICAL TRIAL: NCT07401992
Title: Effects of Semaglutide on Clinical Outcomes and Metabolic Inflammation in Psoriasis: A Randomized, Triple-Blind, Placebo-Controlled Clinical Trial
Brief Title: Effects of Semaglutide on Clinical Outcomes and Metabolic Inflammation in Psoriasis
Acronym: SEMAPSO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Jorge Valdespino Valdes, MD, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DE26-00001
Record Dates: First submitted 2026-01-27; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Psoriasis (PsO); Obesity & Overweight; Diabetes Mellitus - Type 2
Keywords: clinical trial; psoriasis; dermatology; semaglutide; GLP-1; obesity; overweight; diabetes
MeSH Terms: conditions — Psoriasis; Obesity; Overweight; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide group (Active Comparator): A total of 31 participants will be randomly assigned to the semaglutide intervention group.
  Interventions: Drug: Semaglutide (Rybelsus®)
- Placebo group (Placebo Comparator): A total of 31 participants will be randomly assigned to the placebo intervention group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide (Rybelsus®) — Oral semaglutide will be administered once daily at a dose of 3 mg for the first 4 weeks, followed by 7 mg once daily for the next 4 weeks, and 14 mg once daily for the final 4 weeks (total treatment duration: 12 weeks). All participants will also receive conventional topical therapy for 12 weeks, consisting of a topical corticosteroid and a vitamin D analog (calcipotriol).
  Arms: Semaglutide group
Drug: Placebo — A total of 31 participants will be randomly assigned to the placebo intervention group. They will receive a daily placebo tablet containing starch for 12 weeks. All participants will also receive conventional topical therapy for 12 weeks, consisting of a topical corticosteroid and a vitamin D analog (calcipotriol).
  Arms: Placebo group

SUMMARY:
This study will evaluate the effects of oral semaglutide in combination with topical corticosteroid/calcipotriol on clinical outcomes and metabolic inflammation in patients with plaque psoriasis and overweight/obesity and/or type 2 diabetes mellitus. A total of 62 participants will be randomized to receive either semaglutide plus topical corticosteroid/calcipotriol or placebo plus topical corticosteroid/calcipotriol for 12 weeks. Clinical efficacy will be assessed using the Psoriasis Area and Severity Index (PASI), and quality of life will be evaluated using DLQI, PROMIS-29, and EQ-5D-5L. Systemic inflammatory markers will also be measured to assess metabolic inflammation.

DETAILED DESCRIPTION:
Psoriasis is a chronic inflammatory skin disease frequently associated with metabolic comorbidities, including obesity and type 2 diabetes mellitus. Increasing evidence suggests that systemic metabolic inflammation may contribute to psoriasis severity and treatment response. Semaglutide, a glucagon-like peptide-1 (GLP-1) receptor agonist widely used in the management of type 2 diabetes and obesity, has demonstrated anti-inflammatory effects that may be relevant to psoriasis.

This study is a randomized, triple-blind, placebo-controlled clinical trial designed to evaluate the effects of oral semaglutide on clinical disease activity, quality of life, and metabolic inflammatory markers in patients with plaque psoriasis and overweight/obesity and/or type 2 diabetes mellitus.

A total of 62 participants will be enrolled and randomized in a 1:1 ratio to one of two treatment groups. One group will receive oral semaglutide in combination with topical corticosteroid/calcipotriol cream, while the comparator group will receive oral placebo in combination with topical corticosteroid/calcipotriol cream. All participants will receive treatment for 12 weeks.

Clinical assessments will be performed at baseline and at weeks 4, 8, and 12. Disease severity and clinical response will be evaluated using the Psoriasis Area and Severity Index (PASI) at each visit. Patient-reported quality of life will be assessed using the Dermatology Life Quality Index (DLQI), the Patient-Reported Outcomes Measurement Information System-29 (PROMIS-29), and the EuroQol 5-Dimension 5-Level questionnaire (EQ-5D-5L) at baseline and at week 12.

Blood samples will be collected at baseline and at week 12 to evaluate systemic inflammatory and metabolic biomarkers, allowing assessment of changes in metabolic inflammation associated with treatment.

The primary hypothesis is that participants receiving semaglutide in combination with topical corticosteroid/calcipotriol will demonstrate greater improvement in clinical severity and inflammatory markers compared with those receiving placebo plus topical corticosteroid/calcipotriol. Findings from this study may provide evidence supporting the role of metabolic-targeted therapies as adjunctive treatment in psoriasis patients with metabolic comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged ≥18 years at the time of randomization.
* Clinical diagnosis of plaque psoriasis with Psoriasis Area and Severity Index (PASI) ≥3 and body surface area (BSA) ≥3%.
* Body mass index (BMI) ≥25 kg/m², consistent with overweight or obesity.
* Participants with or without type 2 diabetes mellitus.
* Participants with diabetes must be on stable antidiabetic therapy (no changes in medication or dosage within the previous 3 months) and have adequate glycemic control, defined as HbA1c ≤9.0% at baseline.
* No use of systemic psoriasis therapies (e.g., methotrexate, cyclosporine) for at least 8 weeks prior to randomization.
* No use of biologic therapies for at least 3 months prior to randomization.

Exclusion Criteria:

* Diagnosis of a non-plaque psoriasis subtype, including pustular, guttate, nail, inverse, psoriatic arthritis, or erythrodermic psoriasis.
* Pregnancy or breastfeeding at the time of screening or enrollment.
* Insulin-dependent diabetes mellitus or current use of sulfonylureas.
* Active malignancy at the time of screening.
* History of thyroid neoplasia.
* Presence of autoimmune diseases.
* Use of systemic therapies within 8 weeks prior to randomization.
* Use of biologic therapies within 3 months prior to randomization.
* Renal insufficiency.
* Heart failure.
* Hepatic insufficiency.
* History of pancreatitis.
* Current treatment with other GLP-1 receptor agonists.
* History of inflammatory bowel disease.
* Known allergy to starch.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Effect of GLP-1 Receptor Agonists on SCD-1 Activity | Baseline to Week 12
  Change in SCD-1 activity, assessed via acylcarnitine profile (µmol/L), from baseline to Week 12.

SECONDARY OUTCOMES:
Proportion of Participants Achieving Psoriasis Area and Severity Index (PASI) 75 | Weeks 4, 8, and 12
  The proportion of participants achieving a 75% reduction from baseline in the Psoriasis Area and Severity Index (PASI 75) will be compared between the semaglutide and placebo groups.
  The Psoriasis Area and Severity Index (PASI) is a validated clinical severity score that ranges from 0 to 72, with higher scores indicating more severe psoriasis. Achievement of PASI 75 represents a clinically meaningful improvement in disease severity.
Change in Body Weight | Baseline and Week 12
  Change in body weight (kilograms) from baseline to Week 12 will be compared between the semaglutide and placebo groups.
Change in Fasting Plasma Glucose | Baseline and Week 12
  Change in fasting plasma glucose (mg/dL) from baseline to Week 12 will be compared between the semaglutide and placebo groups.
Change in Total Cholesterol | Baseline and Week 12
  Change in serum total cholesterol (mg/dL) from baseline to Week 12 will be compared between the semaglutide and placebo groups.
Correlation Between Metabolic Parameters and PASI Improvement | Baseline to Week 12
  Correlations between PASI improvement and glycemic control (fasting plasma glucose, HbA1c), lipid profile, and anthropometric and hemodynamic parameters (body weight, BMI, waist circumference, hip circumference, waist-to-hip ratio, and blood pressure) will be evaluated overall and by treatment group.
Change in Dermatology Life Quality Index (DLQI) | Baseline and Week 12
  Change from baseline to Week 12 in the Dermatology Life Quality Index (DLQI) score will be compared between the semaglutide and placebo groups.
  The Dermatology Life Quality Index (DLQI) is a validated dermatology-specific quality-of-life questionnaire consisting of 10 items, with total scores ranging from 0 to 30, where higher scores indicate greater impairment in quality of life.
Correlation Between Psoriasis Severity and Quality of Life Measures | Baseline to Week 12
  The correlation between psoriasis severity, measured by the Psoriasis Area and Severity Index (PASI), and quality of life, measured by the Dermatology Life Quality Index (DLQI), Patient-Reported Outcomes Measurement Information System 29-Item Profile (PROMIS-29), and EuroQol 5-Dimensions 5-Levels (EQ-5D-5L), will be assessed overall and by treatment group from baseline to Week 12.
  PASI ranges from 0 to 72, with higher scores indicating more severe psoriasis. DLQI ranges from 0 to 30, with higher scores indicating greater quality-of-life impairment. PROMIS-29 domain scores are reported as T-scores (mean 50, SD 10); higher scores indicate worse symptoms for most domains, except physical function and social roles, where higher scores indicate better functioning. EQ-5D-5L index scores typically range from less than 0 to 1.0, with higher scores indicating better health-related quality of life.
Change in Serum Interleukin-6 (IL-6) | Baseline and Week 12
  Change in serum interleukin-6 (IL-6) levels from baseline to Week 12 will be compared between the semaglutide and placebo groups.
Correlation Between PASI and Inflammatory Biomarkers | Baseline to Week 12
  Correlations between PASI scores and serum levels of IL-6, IL-17, IL-23, TNF-α, CRP, and ESR will be evaluated overall and by treatment group.
PASI Response by Type 2 Diabetes Status | Baseline to Week 12
  Improvement in PASI scores and the proportion of participants achieving PASI 75 and PASI 90 will be compared between participants with and without type 2 diabetes mellitus, stratified by treatment group.
Change in Body Weight in Participants with Type 2 Diabetes | Baseline and Week 12
  Change in body weight (kg) from baseline to Week 12 in participants with type 2 diabetes mellitus.
Change in Serum IL-6 by Diabetes Status | Baseline and Week 12
  Change in serum interleukin-6 (IL-6) levels from baseline to Week 12 will be compared between participants with and without type 2 diabetes mellitus to evaluate differences in semaglutide-induced inflammatory modulation.
Correlation Between Baseline Glycemic Control and Change in Psoriasis Severity | Baseline to Week 12
  The correlation between baseline glycemic control, measured by fasting plasma glucose (mg/dL) and glycated hemoglobin (HbA1c, %), and change in psoriasis severity, measured by the Psoriasis Area and Severity Index (PASI), will be assessed overall and by treatment group from baseline to Week 12.
  The Psoriasis Area and Severity Index (PASI) ranges from 0 to 72, with higher scores indicating more severe psoriasis.
Incidence and Type of Adverse Events | Up to Week 12
  Incidence, type, and severity of adverse events associated with semaglutide, reported as number (%) of participants, up to Week 12.
Change in Body Mass Index (BMI) | Baseline and week 12
  Change in body mass index (BMI, kg/m²) from baseline to Week 12 will be compared between the semaglutide and placebo groups.
Change in Waist Circumference | Baseline and Week 12
  Change in waist circumference (centimeters) from baseline to Week 12 will be compared between the semaglutide and placebo groups.
Change in Hip Circumference | Baseline and Week 12
  Change in hip circumference (centimeters) from baseline to Week 12 will be compared between the semaglutide and placebo groups.
Change in Waist-to-Hip Ratio | Baseline and Week 12
  Change in waist-to-hip ratio from baseline to Week 12 will be compared between the semaglutide and placebo groups.
Change in Blood Pressure | Baseline and Week 12
  Change in systolic and diastolic blood pressure (mmHg) from baseline to Week 12 will be compared between the semaglutide and placebo groups.
Time to First Achievement of PASI 75 | Up to Week 12
  Time to first achievement of a 75% reduction from baseline in the Psoriasis Area and Severity Index (PASI 75) will be compared between the semaglutide and placebo groups.
  The Psoriasis Area and Severity Index (PASI) ranges from 0 to 72, with higher scores indicating more severe psoriasis. Shorter time to PASI 75 represents a better clinical outcome.
Change in PROMIS-29 Profile Score | Baseline and Week 12
  Change from baseline to Week 12 in Patient-Reported Outcomes Measurement Information System 29-Item Profile (PROMIS-29) scores will be compared between the semaglutide and placebo groups.
  PROMIS-29 is a validated patient-reported outcome instrument that assesses multiple health domains. Domain scores are reported as T-scores standardized to a mean of 50 and a standard deviation of 10. For most domains, higher scores indicate worse symptoms or greater impairment, except for physical function and social roles, where higher scores indicate better functioning.
Change in EQ-5D-5L Index Score | Baseline and Week 12
  Change from baseline to Week 12 in the EuroQol 5-Dimensions 5-Levels (EQ-5D-5L) index score will be compared between the semaglutide and placebo groups.
  The EQ-5D-5L is a standardized instrument for measuring health-related quality of life. Index scores typically range from less than 0 (health states worse than death) to 1.0, where higher scores indicate better health status.
Change in Serum Interleukin-17 (IL-17) | Baseline and Week 12
  Change in serum interleukin-17 (IL-17) levels from baseline to Week 12 will be compared between the semaglutide and placebo groups.
Change in Serum Interleukin-23 (IL-23) | Baseline and Week 12
  Change in serum interleukin-23 (IL-23) levels from baseline to Week 12 will be compared between the semaglutide and placebo groups.
Change in Serum Tumor Necrosis Factor-Alpha (TNF-α) | Baseline and Week 12
  Change in serum tumor necrosis factor-alpha (TNF-α) levels from baseline to Week 12 will be compared between the semaglutide and placebo groups.
Change in Serum C-Reactive Protein (CRP) | Baseline and Week 12
  Change in serum C-reactive protein (CRP) levels from baseline to Week 12 will be compared between the semaglutide and placebo groups.
Change in Erythrocyte Sedimentation Rate (ESR) | Baseline and Week 12
  Change in erythrocyte sedimentation rate (ESR) from baseline to Week 12 will be compared between the semaglutide and placebo groups.
Correlation Between Baseline Glycemic Control and Change in Metabolic Parameters | Baseline to Week 12
  The correlation between baseline glycemic control, measured by fasting plasma glucose (mg/dL) and glycated hemoglobin (HbA1c, %), and changes in metabolic parameters, including body weight (kg), body mass index (kg/m²), and serum acylcarnitine profile, will be assessed overall and by treatment group from baseline to Week 12.
Change in Body Mass Index (BMI) by Diabetes Status | Baseline and Week 12
  Change in body mass index (BMI, kg/m²) from baseline to Week 12 will be compared between participants with and without type 2 diabetes mellitus.
Change in Acylcarnitine Profile by Diabetes Status | Baseline and Week 12
  Change in serum acylcarnitine profile from baseline to Week 12 will be compared between participants with and without type 2 diabetes mellitus.
Change in Serum IL-17 by Diabetes Status | Baseline and Week 12
  Change in serum interleukin-17 (IL-17) levels from baseline to Week 12 will be compared between participants with and without type 2 diabetes mellitus.
Change in Serum IL-23 by Diabetes Status | Baseline and Week 12
  Change in serum interleukin-23 (IL-23) levels from baseline to Week 12 will be compared between participants with and without type 2 diabetes mellitus.
Change in Serum TNF-α by Diabetes Status | Baseline and Week 12
  Change in serum tumor necrosis factor-alpha (TNF-α) levels from baseline to Week 12 will be compared between participants with and without type 2 diabetes mellitus.
Change in Serum CRP by Diabetes Status | Baseline and Week 12
  Change in serum C-reactive protein (CRP) levels from baseline to Week 12 will be compared between participants with and without type 2 diabetes mellitus.
Change in ESR by Diabetes Status | Baseline and Week 12
  Change in erythrocyte sedimentation rate (ESR) from baseline to Week 12 will be compared between participants with and without type 2 diabetes mellitus.
Change in HbA1c | Baseline to Week 12
  Change in glycated hemoglobin (HbA1c, %) from baseline to Week 12.
Change in HDL Cholesterol | Baseline to Week 12
  Change in HDL cholesterol (mg/dL) from baseline to Week 12 will be compared between the semaglutide and placebo groups.
Change in LDL Cholesterol | Baseline to Week 12
  Change in LDL cholesterol (mg/dL) from baseline to Week 12 will be compared between the semaglutide and placebo groups.
Change in VLDL Cholesterol | Baseline to Week 12
  Change in VLDL cholesterol (mg/dL) from baseline to Week 12 will be compared between the semaglutide and placebo groups.
Change in Triglycerides | Baseline to Week 12
  Change in triglycerides (mg/dL) from baseline to Week 12 will be compared between the semaglutide and placebo groups.
Change in Body Weight in Participants without Type 2 Diabetes | Baseline to Week 12
  Change in body weight (kg) from baseline to Week 12 in participants without type 2 diabetes mellitus.
Change in Body Mass Index (BMI) in Participants with Type 2 Diabetes | Baseline to Week 12
  Change in BMI (kg/m²) from baseline to Week 12 in participants with type 2 diabetes mellitus.
Change in Body Mass Index (BMI) in Participants without Type 2 Diabetes | Baseline to Week 12
  Change in BMI (kg/m²) from baseline to Week 12 in participants without type 2 diabetes mellitus.
Change in Serum IL-6 in Participants with Type 2 Diabetes | Baseline to Week 12
  Change in serum interleukin-6 (IL-6, pg/mL) from baseline to Week 12 in participants with type 2 diabetes mellitus.
Change in Serum IL-6 in Participants without Type 2 Diabetes | Baseline to Week 12
  Change in serum interleukin-6 (IL-6, pg/mL) from baseline to Week 12 in participants without type 2 diabetes mellitus.
Change in Serum IL-17 in Participants without Type 2 Diabetes | Baseline to Week 12
  Change in serum interleukin-17 (IL-17, pg/mL) from baseline to Week 12 in participants without type 2 diabetes mellitus.
Change in Serum IL-17 in Participants with Type 2 Diabetes | Baseline to Week 12
  Change in serum interleukin-17 (IL-17, pg/mL) from baseline to Week 12 in participants with type 2 diabetes mellitus.
Change in Serum IL-23 in Participants with Type 2 Diabetes | Baseline to Week 12
  Change in serum interleukin-23 (IL-23, pg/mL) from baseline to Week 12 in participants with type 2 diabetes mellitus.
Change in Serum IL-23 in Participants without Type 2 Diabetes | Baseline to Week 12
  Change in serum interleukin-23 (IL-23, pg/mL) from baseline to Week 12 in participants without type 2 diabetes mellitus.
Change in Serum TNF-α in Participants with Type 2 Diabetes | Baseline to Week 12
  Change in serum tumor necrosis factor-alpha (TNF-α, pg/mL) from baseline to Week 12 in participants with type 2 diabetes mellitus.
Change in Serum TNF-α in Participants without Type 2 Diabetes | Baseline to Week 12
  Change in serum tumor necrosis factor-alpha (TNF-α, pg/mL) from baseline to Week 12 in participants without type 2 diabetes mellitus.
Change in Serum C-Reactive Protein (CRP) in Participants with Type 2 Diabetes | Baseline to Week 12
  Change in serum C-reactive protein (CRP, mg/L) from baseline to Week 12 in participants with type 2 diabetes mellitus.
Change in Serum C-Reactive Protein (CRP) in Participants without Type 2 Diabetes | Baseline to Week 12
  Change in serum C-reactive protein (CRP, mg/L) from baseline to Week 12 in participants without type 2 diabetes mellitus.
Change in Erythrocyte Sedimentation Rate (ESR) in Participants with Type 2 Diabetes | Baseline to Week 12
  Change in erythrocyte sedimentation rate (ESR, mm/h) from baseline to Week 12 in participants with type 2 diabetes mellitus.
Change in Erythrocyte Sedimentation Rate (ESR) in Participants without Type 2 Diabetes | Baseline to Week 12
  Change in erythrocyte sedimentation rate (ESR, mm/h) from baseline to Week 12 in participants without type 2 diabetes mellitus.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Dr. José E. González, Monterrey, N.L., Mexico

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF